CLINICAL TRIAL: NCT01819675
Title: Effect of rTMS Over Primary Motor Cortex on Gamma-aminobutyric Acid A (GABAA)-[18F]Flumazenil Binding: A Positron Emission Tomography (PET) Study
Brief Title: Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) Over the Brain on the Neurotransmitter Binding
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: exposure to radiation due to repetitive PET evaluation
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: E-1211-178-001
Record Dates: First submitted 2013-03-19; First posted 2013-03-27 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Stroke; Hemiplegia
Keywords: Neuronal plasticity; Neurotransmitter agents; Receptors, neurotransmitter; Transcranial magnetic stimulation; Stroke; gamma-Aminobutyric Acid
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High frequency (10Hz) rTMS (Experimental): <high frequency rTMS parameters> Intensity: 120% of resting motor threshold; Location: Motor hotspot in primary motor cortex for the dominant hand; Frequency: 10Hz; Number of total stimuli: 750; Coil orientation: tangential to scalp
  Interventions: Device: High frequency rTMS
- Low frequency (1Hz) rTMS (Experimental): <low frequency rTMS parameters> Intensity: 120% of resting motor threshold; Location: Motor hotspot in primary motor cortex for the dominant hand; Frequency: 1Hz; Number of total stimuli: 1200; Coil orientation: tangential to the scalp
  Interventions: Device: Low frequency rTMS
- Sham rTMS (Sham Comparator): <Sham rTMS parameters> Intensity: 120% of resting motor threshold; Location: Motor hotspot in primary motor cortex for the dominant hand; Frequency: 1Hz; Number of total stimuli: 1200; Coil orientation: perpendicular to scalp
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Low frequency rTMS
  Other Names: Magpro (low frequency)
  Arms: Low frequency (1Hz) rTMS
Device: High frequency rTMS
  Other Names: Magpro (high frequency)
  Arms: High frequency (10Hz) rTMS
Device: Sham rTMS
  Other Names: Magpro (sham)
  Arms: Sham rTMS

SUMMARY:
The purpose of this study is to determine whether repetitive transcranial magnetic stimulation (rTMS) over the brain can modulate the binding of neurotransmitter (GABA in this study) to its receptor using the special PET study.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) can modulate the excitability of cortex but exact mechanism is not well determined in human-beings. Changes in some neurotransmitters' status in brain after rTMS have been suggested as a possible mechanism, but role of GABA is not clear.

Twelve healthy people will be recruited. They will receive the rTMS over the primary motor cortex of the dominant hand. Individual subject will receive three sessions of rTMS with wash-out period (more than 3 days) between the rTMS sessions. Three rTMS sessions are high frequency (10Hz), low frequency (1Hz) and sham rTMS. The order of rTMS sessions will be randomly decided. After completing each rTMS session, [18F]flumazenil-PET will be checked.

The purpose of this study is to investigate 1)whether rTMS over the primary motor cortex can modulate the [18F]flumazenil binding potential and 2)whether the modulation of [18F]flumazenil binding potential by rTMS can be different according to the applied frequency of rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people
* 18-50 yrs old
* Right handedness
* Written informed consent

Exclusion Criteria:

* Previous medical diseases such as seizure, stroke, diabetes, hypertension.
* Taking any drugs
* Smoker
* Pregnancy
* Contraindication of PET or MRI
* Stroke or any tumor in MRI
* Metals objects in the head or eyes
* Cardiac pacemaker or cochlear implant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
[18F]flumazenil binding potential | up to 3 months
  Immediately after rTMS session , PET image will be acquired. By using these images, [18F]flumazenil binding potential will be calculated in selected anatomical region up to 3 months

SECONDARY OUTCOMES:
Purdue pegboard test score | Before rTMS (baseline) and average 2hours after rTMS
  evaluation for hand function

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, MD, PhD, Principal Investigator — Department of Rehabilitation Medicine, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam, Korea
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Ayache SS, Farhat WH, Zouari HG, Hosseini H, Mylius V, Lefaucheur JP. Stroke rehabilitation using noninvasive cortical stimulation: motor deficit. Expert Rev Neurother. 2012 Aug;12(8):949-72. doi: 10.1586/ern.12.83. PMID 23002939
- [Background] Malenka RC, Bear MF. LTP and LTD: an embarrassment of riches. Neuron. 2004 Sep 30;44(1):5-21. doi: 10.1016/j.neuron.2004.09.012. PMID 15450156
- [Background] Thickbroom GW. Transcranial magnetic stimulation and synaptic plasticity: experimental framework and human models. Exp Brain Res. 2007 Jul;180(4):583-93. doi: 10.1007/s00221-007-0991-3. Epub 2007 Jun 12. PMID 17562028
- [Background] Yue L, Xiao-lin H, Tao S. The effects of chronic repetitive transcranial magnetic stimulation on glutamate and gamma-aminobutyric acid in rat brain. Brain Res. 2009 Mar 13;1260:94-9. doi: 10.1016/j.brainres.2009.01.009. Epub 2009 Jan 12. PMID 19401169
- [Background] Trippe J, Mix A, Aydin-Abidin S, Funke K, Benali A. theta burst and conventional low-frequency rTMS differentially affect GABAergic neurotransmission in the rat cortex. Exp Brain Res. 2009 Dec;199(3-4):411-21. doi: 10.1007/s00221-009-1961-8. PMID 19701632